CLINICAL TRIAL: NCT04295473
Title: Comparison the Short and Long-term Outcome of Patients With Gastric Cancer Who Underwent Reduced Port Laparoscopic Gastrectomy With Patients Underwent Traditional Laparoscopic Gastrectomy
Brief Title: Reduced Port Laparoscopic Gastrectomy for Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Responsible Party: Principal Investigator, Yunhong Tian, Professor, Nanchong Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020002
Record Dates: First submitted 2020-02-29; First posted 2020-03-04 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Laparoscopic; Gastrectomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced port laparoscopic gastrectomy (Experimental): The definition of reduced port laparoscopic gastrectomy was 1-3 ports used in laparoscopic gastrectomy for gastric cancer.
  Interventions: Procedure: Reduced port laparoscopic gastrectomy
- Standard laparoscopic gastrectomy (No Intervention): 5 ports were used in standard laparoscopic gastrectomy

INTERVENTIONS:
Procedure: Reduced port laparoscopic gastrectomy — The ports were reduced in the surgery of intervention arm.
  Arms: Reduced port laparoscopic gastrectomy

SUMMARY:
Reduced port laparoscopic gastrectomy has been adopted in clinical. The safety and outcome of reduced port laparoscopic gastrectomy has not been systematically evaluated. The investigators sought to compare the short and long-term outcome of patients with gastric cancer who underwent reduced port gastrectomy with patients underwent traditional laparoscopic gastrectomy

DETAILED DESCRIPTION:
Reduced port laparoscopic gastrectomy has been adopted in clinical. The safety and outcome of reduced port laparoscopic gastrectomy has not been systematically evaluated. The investigators designed a comparative study, which sought to compare the short and long-term outcome of patients with gastric cancer who underwent reduced port gastrectomy with patients underwent traditional laparoscopic gastrectomy. The short-term outcome include surgical complications, postoperative morbidity, postoperative nutrition. The long-term outcome mainly include long-term survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the stomach, T1-T4 stages.
2. Eastern Cooperative Oncology Group performance status of 0 or 1.
3. Adequate organ function.

Exclusion Criteria:

1. Patients had distant metastasis.
2. oesophageal invasion of more than 3 cm.
3. Borrmann type 4 or large (more than 8 cm) type 3 carcinoma.
4. Previous chemotherapy or radiation therapy for any other malignancies.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
5-year survival rate | 5 years
  Longterm survival for patients with gastrectomy after reduced port laparoscopic gastrectomy
3-year survival rate | 3 years
  Survival rate for patients with gastrectomy after reduced port laparoscopic gastrectomy

SECONDARY OUTCOMES:
Postoperative morbidity rate | 6 months
  Postoperative morbidity rate for patients with gastrectomy after reduced port laparoscopic gastrectomy
Malnutrition rate | 6 months
  Malnutrition rate for patients with gastrectomy after reduced port
Quality of life in PGSAS-45 scale | 12 months
  The quality of life were assessed using PGSAS-45 scale for patients with gastrectomy after reduced port laparoscopic gastrectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Yunhong Tian, MD, Principal Investigator — Nanchong Central Hospital
Locations (1):
- Yunhong Tian, Nanchong, Sichuan, China